CLINICAL TRIAL: NCT04987086
Title: A Single Center Prospective Study of Diagnostic Efficiency of 68Ga-PSMA PET in the Patients With Locally Advanced and Advanced Renal Cell Carcinoma
Brief Title: 68Ga-PSMA PET in the Renal Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Qin Weijun, Professor and Director, Department of Urology, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20212033-F-1
Record Dates: First submitted 2021-07-11; First posted 2021-08-03 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Renal Cancer; Metastases; PSMA PET
Keywords: advnaced renal cancer; PSMA PET; metastases
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSMA PET Arm (Experimental): The PSMA PET arm received PSMA PET and enhanced CT at the same time in the diagnosis of the patients with suspected renal cancer.
  Interventions: Diagnostic Test: PSMA PET

INTERVENTIONS:
Diagnostic Test: PSMA PET — PSMA PET may have influence on the clinical decision-making of the patients with renal cancer

SUMMARY:
The primary research purpose is to evaluate the diagnostic efficacy of 68Ga-PSMA PET in metastatic lesions of locally advanced and advanced renal cell carcinoma, and to compare with that of enhanced CT. The second purpose is to evaluate whether 68Ga-PSMA PET can change the treatment decision of patients with locally advanced and advanced renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* 2017 AJCC renal cell carcinoma TNM stage III, IV lesions;
* In contrast-enhanced CT staging, suspicious metastases were found;
* There were no known peripheral or central venous problems;
* 68Ga PSMA PET / CT imaging can be performed within 6 weeks after the diagnosis of renal cell carcinoma;
* Signed the informed consent form of voluntary participation in clinical trials.

Exclusion Criteria:

* Age ≤ 18 years old;
* Can't stand lying flat in PET / CT examination;
* There are contraindications for 68Ga PSMA ligands;
* In the past two years, there was a history of other malignant tumors, or according to the doctor's research judgment, complications may occur and affect the normal operation of the test;
* Renal function is impaired or hemodialysis is in progress.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Additional diagnostic value of 68Ga PSMA PET / CT compared with CT in patients with locally advanced and advanced renal cell carcinoma | 2 years
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 68Ga-PSMA PET/CT compared with enhanced CT in diagnosing locally advanced and advanced renal cell carcinoma metastases in clinical practice. If the diagnostic performance of 68Ga PSMA PET / CT is better than enhanced CT, it may have additional diagnostic value in in locally advanced and advanced renal cell carcinoma.

SECONDARY OUTCOMES:
The changes of treatment decision-making in patients with locally advanced and advanced renal cell carcinoma by 68Ga PSMA PET / CT. | 2 years
  The impact of 68Ga-PSMA PET/CT on clinical decisions in patients with locally advanced (Stage III) and advanced renal cell carcinoma (Stage IV) were evaluated by a multidisciplinary prostate cancer therapy team. The clinical decisions were made according to the EAU and NCCN guidelines. The patients with locally advanced (Stage III) has no metastases and advanced renal cell carcinoma (Stage IV) may have oligometastatic disease or metastatic disease. For the patients with locally advanced renal cell carcinoma (Stage III), radical nephrectomy or partial nephrectomy is appropriate. For the patients with advanced renal cell carcinoma (Stage IV), the patients with potentially surgically resectable RCC can receive surgery and the patients with unresectable RCC need to receive systemic therapy and rediotherapy. The different staging performance of enhanced CT and 68Ga-PSMA PET/CT may have impact on patients with locally advanced and advanced renal cell carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaan'xi, China

IPD SHARING:
Plan to Share IPD: No